CLINICAL TRIAL: NCT06252233
Title: Improvement of Quality of Life (QoL) Using Preference-Oriented QoLMonitoring and Linkage with Clinical Registry Data: Randomised Clinical Trial in Patients with Lung Cancer
Brief Title: Improvement of Quality of Life (QoL) Using Preference-Oriented QoLMonitoring in Patients with Lung Cancer
Acronym: LePaLuMo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bayreuth (Other)
Collaborators: University of Regensburg, Tumor Center Regensburg, Center for Quality Management and Health Services Research (Unknown); G-BA Innovationsfonds (Unknown); University Hospital Regensburg, Center for Clinical Trials (Unknown); Bavarian Cancer Registry, Bavarian Health and Food Safety Authority (Unknown)
Responsible Party: Principal Investigator, Martin Emmert, Prof. Dr. Martin Emmert, University of Bayreuth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LePaLuMo_2023
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer; Quality of Life
Keywords: quality of life; lung cancer; definitive randomised controlled trial; patient empowerment; quality of life monitoring; patient and physician preferences
MeSH Terms: conditions — Lung Neoplasms; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient- and physician-centered QoL monitoring (Experimental): Quality of life (QoL) of patients is assessed with an electronic patient- and physician-centered QoL monitoring system using the questionnaires EORTC QLQ-C30 and QLQ-LC29 at study entry and at 1, 2, 3, 4, 5, and 6 months during follow-up care. Results of QoL monitoring are automatically transferred to a QoL profile. Patients and their treating physicians receive the results of their QoL monitoring in real-time. In order to be able to treat QoL deficits a multiprofessional network of therapists is established (e.g. pain therapy, psychotherapy, social support, nutrition counselling, physiotherapy, fitness, respiratory therapy). Intervention group physicians and patients receive complete lists of QoL healthcare professionals of this network practicing in their region. To provide continuous medical education, quality circles for therapy options have been founded.
  Interventions: Behavioral: patient- and physician-centered QoL monitoring
- Routine care (Placebo Comparator): QoL of patients is also assessed with the same QoL monitoring system used in the intervention group at study entry and at 1, 2, 3, 4, 5, and 6 months but neither patients nor treating physicians have access to the QoL profiles. The therapist network is also available for control arm.
  Interventions: Other: Placebo

INTERVENTIONS:
Behavioral: patient- and physician-centered QoL monitoring — Electronic QoL monitoring including QoL diagnosis and therapy (pain therapy, psychotherapy, social support, nutrition, physiotherapy, fitness, respiratory counselling, palliative care). Patients and treating physicians have access to the results of their QoL monitoring and to a network of local healthcare providers.
  Arms: Patient- and physician-centered QoL monitoring
Other: Placebo — Electronic QoL monitoring without QoL diagnosis and therapy. Patients and treating physicians have no access to the results of their QoL monitoring. The therapist network is also available for control arm.
  Arms: Routine care

SUMMARY:
The purpose of the study is to determine whether a preference-oriented quality of life monitoring with defined diagnostic and therapeutic options improves quality of life in patients with lung cancer during routine follow-up care.

DETAILED DESCRIPTION:
A pathway with quality of life (QoL) diagnosis and therapeutic options for patients with breast cancer and colorectal cancer has been successfully designed, implemented, and evaluated as guided by the Medical Research Council framework for developing and testing complex interventions. In two randomised controlled trials the investigators could demonstrate that patients with breast cancer and colorectal cancer had a benefit from the diagnosis of QoL deficits and tailored therapeutic options in their treatment in terms of a decrease in QoL deficits.

The next step is to extend usability of the QoL system so that it can be as well used by patients with other cancer diagnoses and in other study regions. Therefore, QoL will be assessed using an electronic patient- and physician-centered QoL monitoring system which is based on previous work of the research group. The QoL monitoring system is adapted based on results of a preliminary study using discrete choice experiments (DCE) identifying preferences of lung cancer patients and their physicians regarding the importance of individual QoL dimensions.

In this two-arm randomised, controlled, prospective, pragmatic, multicentre clinical trial with one intervention group and one control group QoL of primary lung cancer patients will be assessed with an electronic patient- and physician-centered QoL monitoring system using the quality of life questionnaires (QLQ) of the European Organisation for Research and Treatment of Cancer EORTC QLQ-C30 (core module) and QLQ-LC29 (lung cancer module) at study entry and at 1, 2, 3, 4, 5, and 6 months during follow-up care. Data of each patient's QoL will be linked with clinical data from the Bavarian Cancer Registry for the purpose of data analysis.

In the intervention group results of QoL monitoring are automatically transferred to a preference-based QoL profile including 8 dimensions on scales of 0-100 (cutoff of a "need for QoL therapy" <50). Patients and their treating physicians receive the results of their QoL monitoring in real-time. In order to be able to treat QoL deficits a multi-professional network of therapists is established (e.g. pain therapy, psychotherapy, social support, nutrition counselling, physiotherapy, fitness, respiratory therapy, palliative care). In the intervention group patients and their physicians receive complete lists of QoL healthcare professionals of this network practicing in their region.

In the control group QoL is also measured but neither patients nor treating physicians have access to the results of QoL monitoring, but the therapist network is also available for this study arm.

The investigators expect that the proportion of patients in both groups with a need for QoL therapy (<50 points in at least one dimension of the QoL profile) will be lower in intervention group patients compared with control group patients at the primary endpoint 6 months after study entry.

ELIGIBILITY:
Inclusion Criteria:

1. primary diagnosis of lung cancer (ICD C33/C34, all stages)
2. treatment in one of six recruiting hospitals treating patients with lung cancer (University Hospital Regensburg, Hospital Barmherzige Brüder Regensburg, Hospital Bayreuth, Hospital Coburg, Hospital Kulmbach, Hospital Bamberg);
3. difference between date of histology and date of study entry not exceeding 2 months;
4. informed consent;

Exclusion Criteria:

1. unavailability of a study clinician for patient recruitment;
2. patient misclassified in the candidate list (no primary diagnosis, no lung tumour);
3. coordinating practitioner refuses trial participation;
4. patient outside the defined study region (Germany, Bavaria: Upper Palatinate, Lower Bavaria, Upper Franconia);
5. age under 18 years;
6. pregnancy/ breastfeeding;
7. patient unable to fill out the QoL questionnaire (physical, psychological, cognitive, language reasons);
8. patient refuses trial participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a need for QoL therapy in at least one dimension of the QoL profile at 6 months | 6 months after study entry
  proportion of patients in both groups with a need for QoL therapy (<50 points) in at least one of eight dimensions of the QoL profile: global quality of life, shortness of breath, physical functioning, social functioning, fear of progression, emotional functioning, pain, financial impact

SECONDARY OUTCOMES:
Proportion of patients with a need for QoL therapy in each dimension of the QoL profile at 1, 2, 3, 4, 5, and 6 months | 1, 2, 3, 4, 5, 6 months after study entry
  proportions of patients with a need for QoL therapy (<50 points) in each single dimension of the QoL profile: global quality of life, shortness of breath, physical functioning, social functioning, fear of progression, emotional functioning, pain, financial impact

CONTACTS AND LOCATIONS:
Overall Officials: Martin Emmert, PhD, Prof., Study Chair — University of Bayreuth, Faculty of Law, Business and Economics, Institute for Healthcare Management and Health Sciences; Monika Klinkhammer-Schalke, MD, Prof., Study Chair — University of Regensburg, Centre for Quality Management and Health Services Resarch
Locations (8):
- Germany (8):
  - Klinikum Bamberg, Bamberg
  - Hospital Bayreuth, Bayreuth
  - Klinikum Coburg GmbH, Coburg
  - Caritas Krankenhaus St. Maria Donaustauf, Donaustauf
  - Klinikum Kulmbach, Kulmbach
  - Krankenhaus Barmherzige Brüder, Regensburg
  - Universitätsklinikum Regensburg, Regensburg
  - Klinikum St. Elisabeth Straubing, Straubing

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data (IPD) that underlie the results in a publication are planned to be made available upon request of scientists.
Supporting Information: Study Protocol
Time Frame: 6 months after date of publication until 60 months after date of publication
Access Criteria: Data will be made available to other scientists upon request for nonprofit research. The contact address is monika.klinkhammer-schalke@ur.de. Scientists are required to send their predefined statistical analysis plan. Together with the scientific review board of the Tumor Center Regensburg a decision will be made based on the quality and usefulness of planned statistical analysis. In case of a positive decision the scientist is required to sign a contract for data usage before receiving anonymized IPD.

REFERENCES:
- [Background] Klinkhammer-Schalke M, Steinger B, Koller M, Zeman F, Furst A, Gumpp J, Obermaier R, Piso P, Lindberg-Scharf P; Regensburg QoL Study Group. Diagnosing deficits in quality of life and providing tailored therapeutic options: Results of a randomised trial in 220 patients with colorectal cancer. Eur J Cancer. 2020 May;130:102-113. doi: 10.1016/j.ejca.2020.01.025. Epub 2020 Mar 13. PMID 32179445
- [Background] Klinkhammer-Schalke M, Koller M, Steinger B, Ehret C, Ernst B, Wyatt JC, Hofstadter F, Lorenz W; Regensburg QoL Study Group. Direct improvement of quality of life using a tailored quality of life diagnosis and therapy pathway: randomised trial in 200 women with breast cancer. Br J Cancer. 2012 Feb 28;106(5):826-38. doi: 10.1038/bjc.2012.4. Epub 2012 Feb 7. PMID 22315052
- [Background] Lindberg-Scharf P, Steinger B, Koller M, Hofstadter A, Ortmann O, Kurz J, Sasse J, Klinkhammer-Schalke M. Long-term improvement of quality of life in patients with breast cancer: supporting patient-physician communication by an electronic tool for inpatient and outpatient care. Support Care Cancer. 2021 Dec;29(12):7865-7875. doi: 10.1007/s00520-021-06270-1. Epub 2021 Jun 27. PMID 34176020
- [Derived] Lindberg-Scharf P, Emmert M, Koller M, Gurtler F, Steinger B, Muller-Nordhorn J, Zeman F, Friebel S, Ibler K, Kurz J, Stangl T, Klinkhammer-Schalke M, Volkel V. Preference-oriented quality of life monitoring and linkage with clinical registry data: study protocol of a randomised clinical trial in patients with lung cancer (LePaLuMo Study). Trials. 2025 Sep 16;26(1):339. doi: 10.1186/s13063-025-09102-3. PMID 40958112